CLINICAL TRIAL: NCT06376474
Title: To Evaluate the Pharmacokinetics of Hemay005 Tablets in Subjects With Mild, Moderate Liver Impairment and Normal Liver Function After a Single Oral Administration
Brief Title: To Evaluate the Pharmacokinetics of Hemay005 Tablets in Subjects With Liver Damage
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM005PS1S06
Record Dates: First submitted 2024-04-09; First posted 2024-04-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Hemay005

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild liver damage group (Experimental): 15mg/tablet，Four tablets (60mg) each time. Participants will receive a single dose of Hemay005 tablet in Day1
  Interventions: Drug: Hemay005
- Moderate liver damage group (Experimental): 15mg/tablet，Four tablets (60mg) each time. Participants will receive a single dose of Hemay005 tablet in Day1
  Interventions: Drug: Hemay005
- Healthy subjects (Experimental): 15mg/tablet，Four tablets (60mg) each time. Participants will receive a single dose of Hemay005 tablet in Day1
  Interventions: Drug: Hemay005

INTERVENTIONS:
Drug: Hemay005 — 15mg/tablet，Four tablets (60mg) each time. Participants will receive a single dose of Hemay005 tablet in Day1
  Other Names: Hemay005 tablet

SUMMARY:
The purpose of this study was to evaluate the pharmacokinetics of Hemay 005 tablets in subjects with mild, moderate liver impairment and normal liver function, and to provide a basis for the formulation of clinical medication regimens for patients with liver impairment.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetics and safety of Hemay 005 tablets in subjects with mild, moderate liver impairment and normal liver function, and to provide a basis for the formulation of clinical medication regimens for patients with liver impairment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Fully understand the content, process and possible adverse reactions of the trial before the trial, and be able to complete the study and sign the informed consent according to the requirements of the trial protocol;

  2. Adults of both sexes aged from 18 to 70 years old (both ends, based on written informed consent);

  3. The body weight of male subjects should not be less than 50 kg and the body weight of female subjects should not be less than 45 kg. Body mass index (BMI) : 19-32 kg/m2 (including cut-off value);

  4. chronic stable liver impairment (no clinically significant change in disease status as judged by the investigator to have occurred for at least 28 days (or up to 14 days for patients with moderate liver function) before taking the study drug) due to primary liver disease (e.g., autoimmune hepatitis, nonalcoholic fatty liver disease, alcoholic liver disease, etc.); Patients were classified as grade A/mild (Child-Pugh score: 5-6) or grade B/moderate (Child-Pugh score: 7-9) according to the Child-Pugh classification within 72 hours before taking the study drug; Among them, the researchers used standard diagnosis and treatment methods, combined with the patient's past medical history, laboratory tests, liver biopsy or imaging examination and other documents to diagnose chronic liver function impairment, and then evaluated according to the Child-Pugh classification.

  5. (Inquiry) patients who have a stable medication plan for the treatment of liver function impairment, complications, and other concomitant diseases for at least 28 days (or 14 days for patients with moderate liver function) before taking the study drug, and who do not need to adjust the medication (including the type, dose, or frequency of medication); Or those who do not use drugs;

  6.In addition to liver function damage and complications, the investigators were in good physical condition according to medical history inquiry, vital signs, physical examination, laboratory tests (blood routine, urine routine, stool routine, blood biochemistry, coagulation function, blood pregnancy (only female), 12-lead electrocardiogram, chest X-ray, abdominal color Doppler ultrasound, electroencephalogram, etc.), and no other clinically significant abnormalities.

Exclusion Criteria:

* 1. (Inquiry) The subject has any of the following conditions: previous liver transplantation; Severe portal hypertension or transsurgical portosystemic shunt; Patients with suspected or confirmed liver cancer or other malignant tumors; Patients with hepatorenal syndrome; Biliary cirrhosis, biliary obstruction, cholestatic liver disease and other diseases that seriously affect bile excretion; Patients with complications such as hepatic encephalopathy (according to Child-Pugh criteria), liver failure, esophageal and gastric varices bleeding, severe/advanced ascites or pleural effusion requiring puncture drainage and albumin supplementation, who were considered by the investigator to be unsuitable;

  2. (Inquiry) In addition to the disease causing liver function impairment, patients with serious acute or chronic diseases of other important organs within 1 year before screening, including but not limited to neuropsychiatric, gastrointestinal, respiratory, urinary, endocrine, hematological, immune and other diseases, judged by the investigator to be not suitable for the trial;

  3. (Inquiry) Any of the following occurred within 6 months prior to study entry: Myocardial infarction, Congenital long QT syndrome, Torsades de pointes (including sustained ventricular tachycardia and ventricular fibrillation), right bundle branch block and left anterior hemiblock (bifascicular block), Unstable angina pectoris, coronary artery/peripheral artery bypass grafting, New York Heart Association (NYHA) class III or IV congestive heart failure, cerebrovascular accident, transient ischemic attack, or pulmonary embolism;

  4. (asking) a history of depression or suicidal tendencies;

  5. (Inquiry) patients who had severe gastrointestinal diseases (except secondary gastrointestinal diseases caused by hepatitis) or had digestive system surgery within 3 months before screening, and the investigators thought that the absorption of drugs was affected;

  6. (Inquiry) patients who lost blood or donated more than 400mL of blood within one month before screening, or received red blood cell transfusion;

  7. (Inquiry) Liver function fluctuation (e.g., active hepatitis), rapid deterioration (e.g., advanced ascites, fever, active gastrointestinal bleeding), CTCAE 5.0 common adverse event grade ≥ 2, ongoing arrhythmia, atrial fibrillation of any grade during screening;

  8.The screening laboratory test results met any of the following: (a) alanine aminotransferase (ALT) >5 times the normal value; (b) neutrophil count <1.0×109/L; (c) hemoglobin (HGB) <90 g/L; (d) platelet level <50×109/L; (e) subjects with alpha-fetoprotein (AFP) >50 ng/mL and suspected hepatocellular carcinoma;

  9. (Inquiry) patients with specific allergic history (asthma, urticaria, eczema, etc.), or allergic condition (such as allergic to two or more drugs, foods or pollens), or known allergic to PDE4 inhibitors (such as apast, roflumilast, etc.);

  10. (inquiry) those who had a history of drug abuse in the past 5 years or drug abuse in the past 3 years before screening;

  11. Screen-positive for drug abuse (except those screen-positive for drug abuse due to concomitant medication);

  12. Positive breath alcohol test (alcohol concentration >0mg/L);

  13. (Inquiry) who consumed more than 14 units of alcohol per week in the 3 months before screening (1 unit = 17.7 mL ethanol, i.e. 1 unit = 354 mL of 5% beer or 44 mL of 40% liquor or 147 mL of 12% wine), or who could not abstain from alcohol during the study;

  14. (Inquiry) who smoked more than 5 cigarettes per day in the 3 months before screening, or who could not stop using any tobacco products during the study;

  15. (Inquiry) subjects who consumed excessive amounts of tea, coffee and/or caffeine-rich beverages (more than 8 cups, 1 cup =250 mL) per day in the previous 3 months;

  16. Having one or more of the tests for hepatitis B, C, HIV and syphilis clinically significant;

  17. (Inquiry) who participated in clinical trials of other drugs/devices within 3 months before screening and used the trial drugs/devices;

  18. (Inquiry) who had received drugs with definite potential hepatotoxicity (such as acetaminophen, statins, azithromycin, dapsone, clarithromycin, fluconazole, ketoconazole, rifampicin, etc.) for 7 consecutive days or more within 3 months before screening;

  19. (Inquiry) Use of any drugs (e.g., inductors-barbiturates, pioglitazone, carbamazepine, phenytoin, glucocorticoids) that induce or inhibit hepatic drug-metabolizing enzymes within 30 days before screening; Inhibitors: SSRI antidepressants, cimetidine, diltiazem macrolides, nitroimidazole, sedative hypnotics, verapamil, fluoroquinolones, antihistamines, isoniazid);

  20. (Inquiry) who used prescription drugs, over-the-counter drugs, health supplements, herbal products or vaccines other than those used for liver function impairment and other concomitant diseases within 2 weeks before screening;

  21. (Inquiry) any caffeine/xanthine/food or drink (such as strong tea, coffee, chocolate, cola, animal organs, grapefruit, dragon fruit, mango, etc.) rich in caffeine/xanthine/may affect the absorption, distribution, metabolism, excretion of drug in the judgment of the investigator during the period from screening to day -1 of admission, or unable to stop the intake of the above food or drink during the trial;

  22. (Asking) pregnant or lactating women, or subjects (including male subjects) who have plans to give birth or donate sperm or eggs from two weeks before the trial to six months after the last dose of drug, unwilling or not to take effective contraceptive measures;

  23. (inquiry) those who are unable to eat or have swallowing difficulties, have special dietary requirements and/or cannot follow a uniform diet;

  24. (inquiry) with a history of epileptic seizures;

  25. (Inquiry) Those who cannot tolerate venipuncture and/or have a history of dizzy with blood and needles;

  26. Subjects with other factors considered by the investigator to be ineligible for the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-28 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Relevant pharmacokinetic parameters，Peak Plasma Concentration（Cmax） | Day1-Day6
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，Area under the plasma concentration versus time curve（AUC0-t） | Day1-Day6
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，Area under the curve from time 0 extrapolated to infinite time (AUC0-inf) | Day1-Day6
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，half-life (T1/2) | Day1-Day6
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，clearance (CL/F) | Day1-Day6
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，volume of distribution (Vz/F) | Day1-Day6
  All subjects who receive the drug will be analyzed for pharmacokinetic

CONTACTS AND LOCATIONS:
Overall Officials: Weiyong Li, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital of Tongji Medical College; Huazhong University of Science and Technology, Wuhan, Hubei, China